CLINICAL TRIAL: NCT02170870
Title: Gastrointestinal Sensorimotor Dysfunctions in Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-002098; P01DK068055 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Dyspepsia; Diabetes Mellitus With Gastrointestinal Symptoms
MeSH Terms: conditions — Dyspepsia | interventions — exendin (9-39); Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Healthy Controls Exendin 9-39 (Experimental): Exendin 9-39 was administered intravenously (1,200 pmol/kg bolus followed by infusion at 300 pmol/kg/min).
  Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Exendin 9-39; Drug: Microlipid
- Healthy Controls Placebo (Placebo Comparator): Normal saline infusion was prepared to match the appearance of Exendin 9-39. Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Microlipid; Drug: Placebo
- Diabetics Exendin 9-39 (Experimental): Exendin 9-39 was administered intravenously (1,200 pmol/kg bolus followed by infusion at 300 pmol/kg/min).
  Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Exendin 9-39; Drug: Microlipid
- Diabetics Placebo (Placebo Comparator): Normal saline infusion was prepared to match the appearance of Exendin 9-39. Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Microlipid; Drug: Placebo
- Functional Dyspepsia Exendin 9-39 (Experimental): Exendin 9-39 was administered intravenously (1,200 pmol/kg bolus followed by infusion at 300 pmol/kg/min).
  Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Exendin 9-39; Drug: Microlipid
- Functional Dyspepsia Placebo (Placebo Comparator): Normal saline infusion was prepared to match the appearance of Exendin 9-39. Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
  Interventions: Drug: Microlipid; Drug: Placebo

INTERVENTIONS:
Drug: Exendin 9-39 — Exendin 9-39 will be administered intravenously (1,200 pmol/kg bolus followed by infusion at 300 pmol/kg/min).
  Arms: Diabetics Exendin 9-39; Functional Dyspepsia Exendin 9-39; Healthy Controls Exendin 9-39
Drug: Microlipid — Lipid infusion {66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
Drug: Placebo — Normal saline infusion will be prepared to match the appearance of Exendin 9-39
  Arms: Diabetics Placebo; Functional Dyspepsia Placebo; Healthy Controls Placebo

SUMMARY:
The purpose of this study is to understand why people with indigestion have gastrointestinal symptoms and in particular to understand whether symptoms are related to increased sensitivity to nutrients in the small intestine and to a hormone (GLP1) which is normally released from the small intestine in response to nutrients. We propose to study the contribution of GLP1 to intestinal sensitivity with a drug (exendin 9-39) that blocks the effects of GLP1.

DETAILED DESCRIPTION:
Upper gastrointestinal symptoms (early satiety, pain, nausea, and vomiting) are not uncommon in diabetic (DM) enteropathy. While these symptoms are often attributed to accelerated or delayed gastric emptying, the precise contribution of abnormal gastric emptying to symptoms in patients with DM gastroparesis is often unclear.

The investigators recently observed that approximately 50% of patients with functional dyspepsia have increased sensation to duodenal nutrient (carbohydrate and lipid) perfusion. Another recent study suggests that patients with functional dyspepsia have low-grade mucosal inflammation, abnormalities of cell-to-cell adhesion proteins which predispose to increased epithelial permeability, and a leaky epithelial barrier. Type 1 DM is associated with increased small intestinal permeability even in subjects who do not have celiac disease.

Hence, the investigators proposed to evaluate the overall hypothesis that intestinal chemosensitivity related to increased epithelial permeability and GLP-1 explains symptom severity in patients with functional dyspepsia and in patients with DM and dyspepsia. Healthy subjects, Patients with DM and GI symptoms, and patients with functional dyspepsia underwent assessment of intestinal chemosensitivity during duodenal nutrient perfusion, gastric emptying (by scintigraphy), cardiovascular and GI vagal functions (plasma pancreatic polypeptide response to sham feeding and a comprehensive autonomic reflex screen), in vivo assessment of small intestinal permeability (urinary lactulose:mannitol ratio), and upper endoscopy with assessment of epithelial tight junction proteins and permeability on small bowel biopsies.

During the nutrient infusion, subjects in each group (i.e., healthy subjects, functional dyspepsia and DM) were randomized to lipid infusion and placebo or lipid infusion and exendin 9-39. Hormonal responses (i.e., GLP-1, cholecystokinin (CCK), gastric inhibitory polypeptide (GIP), glucagon, peptide tyrosine tyrosine (PYY), C-peptide, and insulin) and plasma glucose will also be evaluated during enteral nutrient infusion. GI symptoms during each perturbation (meal, nutrient infusion) will be evaluated by validated questionnaires. Blood will be collected for DNA-based genetic analyses, initially to assess the relationship of GI sensorimotor dysfunctions and symptoms with single nucleotide polymorphisms (SNPs) affecting CCK and GLP-1 receptors. The analysis will assess for disturbances in these parameters in functional and DM dyspepsia, investigate associations between symptoms during enteral infusion and hormonal-epithelial functions, and evaluate relationships between daily symptoms and results of testing.

ELIGIBILITY:
Inclusion criteria for controls:

* Healthy male or non-pregnant, non-breastfeeding female volunteers;
* 18-70 years old;
* Able to provide written informed consent before participating in the study;
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study

Additional inclusion criteria for patients:

* Symptoms of dyspepsia (i.e., early satiety, postprandial discomfort, nausea, vomiting, regurgitation)
* Patients in the Diabetes Mellitus (DM) group will also require Type 1 or 2 DM of ≥ 3 years duration; in patients with type 2 DM, the dyspepsia symptoms should have begun or worsened after DM was diagnosed

Exclusion criteria - for patients and controls:

* Major abdominal surgery (i.e., appendectomy, cholecystectomy, tubal ligation, hysterectomy, and limited colonic resection are permissible)
* Clinical evidence (including physical exam and EKG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Opiates, alpha adrenergic agonists, metoclopramide, and high doses of anticholinergic agents (e.g., amitriptyline greater than 50 mg daily). If medically safe, these drugs may be discontinued for four half lives prior to study assessments
* Treatment with glucagon-like peptide-1 (GLP-1) agonists and amylin which cause vagal blockade and may affect central processing of pain
* Use of tobacco products within the past six months or NSAIDs or aspirin within the past week (since they all may affect intestinal permeability)
* Bleeding or clotting disorders or medications that increase risk of bleeding from mucosal biopsies
* Positive tissue transglutaminase antibodies (TTG)
* For two days prior to studies, subjects will be instructed to avoid ingestion of artificial sweeteners such as sucralose (SplendaTM), aspartame (NutrasweetTM), foods containing lactulose or mannitol
* Pregnant or breast-feeding females
* Known intolerance or allergy to eggs
* Poor peripheral venous access, if central venous access is not available
* Any other condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study

Exclusion criteria for controls only:

• Current symptoms of a functional gastrointestinal disorder assessed by questionnaire

Exclusion criteria for patients only:

* Severe vomiting that would preclude tube placement or participation in the study
* Structural cause for symptoms by endoscopy within the past 48 months
* Patients with gastric pacemakers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-06; Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Chakraborty S, Halland M, Burton D, Desai A, Neja B, Low P, Singer W, Camilleri M, Zinsmeister AR, Bharucha AE. GI Dysfunctions in Diabetic Gastroenteropathy, Their Relationships With Symptoms, and Effects of a GLP-1 Antagonist. J Clin Endocrinol Metab. 2019 Jun 1;104(6):1967-1977. doi: 10.1210/jc.2018-01623. PMID 30358871
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Healthy Controls Exendin 9-39 | Healthy Controls Placebo | Diabetics Exendin 9-39 | Diabetics Placebo | Functional Dyspepsia Exendin 9-39 | Functional Dyspepsia Placebo
Started | 13 | 11 | 20 | 20 | 20 | 20
Completed | 13 | 11 | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls Exendin 9-39 | Healthy Controls Placebo | Diabetics Exendin 9-39 | Diabetics Placebo | Functional Dyspepsia Exendin 9-39 | Functional Dyspepsia Placebo | Total
Number analyzed (Participants) | 13 | 11 | 20 | 20 | 20 | 20 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12.6) | 42 (14.3) | 45 (15.7) | 45 (11.6) | 44 (13.2) | 39 (13) | 42.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 16 | 15 | 15 | 16 | 76
  Male | 5 | 5 | 4 | 5 | 5 | 4 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 20 | 20 | 20 | 20 | 104
BMI [Mean (Standard Deviation); unit: kg/m2] | 26 (4.4) | 26 (5.3) | 29 (6.6) | 27 (4.5) | 26 (6.4) | 27 (6.9) | 26.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Intestinal Chemosensitivity to Lipids Perfusion
Description: Intestinal chemosensitivity was recorded by evaluating symptoms during duodenal lipid infusion (0.5 gm/mL diluted in water to 222 mL) and placebo or the glucagon like peptide 1 (GLP-1) receptor antagonist exendin 9-39 over 2 hours. Participants reported the severity of 6 symptoms (nausea, fullness, bloating, abdominal pain, belching, and burning) at 15 minute intervals using a Visual Analogue Scale (VAS) marked 0 (minimum value) - 4 (maximum value): absent (0), light (1), moderate (2), severe (3) and intolerable(4). The scores recorded for nausea, fullness, bloating, and abdominal pain over the 2 hour infusion were averaged and reported as the mean symptom score. Higher scores mean a worse outcome.
Time Frame: Day 1, approximately 2 hours after infusion
Population: Functional Dyspepsia arm - enteral lipid infusion was not performed because a nasoduodenal tube could not be placed in 2 functional dyspepsia placebo subjects and 3 functional dyspepsia exendin 9-39 subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Controls Exendin 9-39 | Healthy Controls Placebo | Diabetics Exendin 9-39 | Diabetics Placebo | Functional Dyspepsia Exendin 9-39 | Functional Dyspepsia Placebo
Number analyzed (Participants) | 13 | 11 | 20 | 20 | 17 | 18
score on a scale | 0.22 (0.05) | 0.36 (0.13) | 0.55 (0.11) | 0.65 (0.17) | 1.4 (0.9) | 1.2 (0.9)
Statistical Analysis 1: Comparison: Healthy Controls Exendin 9-39 vs Healthy Controls Placebo vs Diabetics Exendin 9-39 vs Diabetics Placebo; Mean GI symptom score during lipid infusion in controls vs diabetics adjusted for treatment status (ie, exendin or placebo); Test type: Superiority; p = 0.06, ANOVA
Statistical Analysis 2: Comparison: Healthy Controls Exendin 9-39 vs Healthy Controls Placebo vs Functional Dyspepsia Exendin 9-39 vs Functional Dyspepsia Placebo; Mean GI symptom score during lipid infusion in controls vs functional dyspepsia adjusted for treatment status (ie, exendin or placebo); Test type: Superiority; p = 0.0001, ANOVA

2. Secondary Outcome: Rate of Gastric Emptying (GE t 1/2) in Patients With Diabetes Mellitus (DM) or Non-ulcer Dyspepsia (NUD) Compared to Placebo
Description: The time for half of the ingested solids or liquids to leave the stomach. Following a meal consisting of two eggs labeled with technetium Tc 99m sulfur colloid (1 mCi) served on one slice of bread with milk labeled with indium In111 diethylenetriaminepentaacetate (0.1 mCi), gastric emptying of solids and liquids was assessed with scintigraphy. Rapid emptying is defined as ≥ 36% emptied at one hour and delayed emptying is defined as < 76% emptied at four hours. Normal emptying is defined as amount less than rapid emptying definition but greater than delayed emptying definition.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Controls; Diabetics Exendin 9-39; Functional Dyspepsia Exendin 9-39: Exendin 9-39 was administered intravenously (1,200 pmol/kg bolus followed by infusion at 300 pmol/kg/min).
  Lipid infusion 66.7 mL Microlipid (0.5 gm/mL diluted in water to 222 ml).
Arm/Group | Healthy Controls | Healthy Controls Placebo | Diabetics Exendin 9-39 | Diabetics Placebo | Functional Dyspepsia Exendin 9-39 | Functional Dyspepsia Placebo
Number analyzed (Participants) | 13 | 11 | 20 | 20 | 20 | 20
Participants
  GE of solids: Rapid emptying | 1 | 3 | 0 | 5 | 2 | 3
  GE of solids: Normal emptying | 10 | 8 | 12 | 10 | 16 | 14
  GE of solids: Delayed emptying | 2 | 0 | 8 | 5 | 2 | 3
  GE of liquids: Rapid emptying | 2 | 2 | 0 | 1 | 1 | 1
  GE of liquids: Normal emptying | 11 | 9 | 19 | 18 | 19 | 19
  GE of liquids: Delayed emptying | 0 | 0 | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: For this study, the study treatment follow-up period was defined as one day following the last administration of study treatment.
Arm/Group | Healthy Controls Exendin 9-39 | Healthy Controls Placebo | Diabetics Exendin 9-39 | Diabetics Placebo | Functional Dyspepsia Exendin 9-39 | Functional Dyspepsia Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 2/20 | 1/20 | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls Exendin 9-39 (N=13) | Healthy Controls Placebo (N=11) | Diabetics Exendin 9-39 (N=20) | Diabetics Placebo (N=20) | Functional Dyspepsia Exendin 9-39 (N=20) | Functional Dyspepsia Placebo (N=20)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02170870/Prot_SAP_000.pdf